CLINICAL TRIAL: NCT04943198
Title: Optimization of the Time and Dosage of Vemurafenib in BRAF Positive Juvenile Patients With Refractory Histiocytosis
Acronym: BRAVO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anna Raciborska (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other); Łukasiewicz Research Network (Unknown); Wrocław University of Environmental and Life Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Anna Raciborska, Prof Ass MD PhD, Institute of Mother and Child, Warsaw, Poland
Organization: Institute of Mother and Child, Warsaw, Poland (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRAVO
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Histiocytosis
Keywords: Langerhans cell histiocytosis (LCH); vemurafenib; children; refractory histiocytosis; paediatric patients
MeSH Terms: conditions — Histiocytosis; Histiocytosis, Langerhans-Cell | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R1 time of vemurafenib treatment (Experimental): vemurafenib will be given to 6 months after BRAF negativization
  Interventions: Drug: Vemurafenib
- R2 time of vemurafenib treatment (Experimental): vemurafenib will be given to 12 months after BRAF negativization
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — 20 mg/kg/day
  Other Names: Zelboraf

SUMMARY:
Prospective, interventional, open, randomized, single-center, non-commercial clinical trial to optimize treatment and dosage of vemurafenib in juvenile patients with histiocytosis resistant to conventional therapy and in whom the BRAF gene mutation has been found.

DETAILED DESCRIPTION:
BRAVO clinical study is part of the POLHISTIO project. The POLHISTIO project is a non-commercial clinical trial aimed at optimizing the diagnosis and treatment of juvenile patients with histiocytosis. The project objectives are defined as follows: 1) to estimate the nature and frequency of mutations in patients with histiocytosis in both tumor tissues and free-circulating DNA; 2) to compare molecular test results with clinical data; 3) to evaluate the diagnostic usefulness of the status of molecular analysis (MRD) as a prognostic factor compared with other recognized factors; 4) in the case of failure of conventional therapy - to modify treatment and to apply targeted treatment, based on molecular status of gene mutation. The project is intended to include patients from all over Poland.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of mutations in the BRAF gene in tumor tissues and/or in circulating tumor DNA (ctDNA) at any stage of treatment or follow-up.
2. Failure of the treatment (at least one of below needs to apply in order for this requirement to be satisfied):

   1. Progression on the I and/or II line treatment, including at least one risk organ; prior treatment should include a minimum of 6 weeks of weekly Vinblastine with a minimum of 28 days prednisolone or minimum 2 cycles of Cytosine Arabinoside in 4-day cycles and/or Cladribine in 5-day cycles as a 2nd line treatment, minimum 2 cycles, or other second-line treatment or
   2. Disease reactivation after an initial response to treatment with Vimblastine and prednisolone as the first line and/or no response to second line treatment using one of two drugs: Cytosine Arabinoside in 4-day cycles and/or Cladribine in 5-day cycles, minimum 2 cycles, or other I/ II line treatment or occurrence of involvement of at least one risk organ or
   3. Third or subsequent reactivation of disease with or without risk organ involvement, or
   4. Reactivation of disease after Vemurafenib therapy has been completed, or
   5. The appearance of signs of neurodegenerative disorder (ND) in MRI of the central nervous system (CNS).
3. Signing of informed consent for trial participation (including for Vemurafenib treatment) according with current legal regulations.
4. Consent to the use of effective contraception throughout the Vemurafenib administration period and a minimum of 1 year after discontinuation in patients at puberty and sexual maturity.
5. Participation in HISTIOGEN trial.

Exclusion Criteria:

1. Lack of inclusion criteria.
2. Pregnancy and breastfeeding .
3. Hypersensitivity to the study drug or any of its ingredients.
4. Iritis, uveitis, obstruction of the retinal veins.
5. Simultaneous treatment with other drugs which might interact with Vemurafenib.
6. Persistent toxicity related to prior therapy, making it impossible to treat with Vemurafenib.
7. Diagnosis of other malignancies before study inclusion.
8. Other acute or persistent disorders, behaviors or abnormal laboratory test results, which might increase the risk related to the participation in this clinical trial or to taking the study drug, or which might influence the interpretation of the study results, or which, in the investigator's opinion, disqualify a patient from participating in the trial.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
event-free survival | 2 years
  Event-free survival (EFS) was defined as the time interval from the date of diagnosis to the date of disease progression, recurrence, second malignancy, death or to date of last follow-up for patients without events.

SECONDARY OUTCOMES:
Molecular relapse (in ct DNA) | 2 years
  Molecular relapse was defined as the time interval from the date of BRAF negativization to the date of positive results of BRAF mutation
Time to negative mutation test results (in ct DNA) | 2 years
  Time to negative mutation test results (in ct DNA) was defined as the time interval from the date of positive BRAF mutation to the date of negative results of BRAF mutation

CONTACTS AND LOCATIONS:
Overall Officials: Anna Raciborska, Principal Investigator — Mother and Child Institute
Locations (1):
- Mother and Child Institute, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badalian-Very G, Vergilio JA, Degar BA, MacConaill LE, Brandner B, Calicchio ML, Kuo FC, Ligon AH, Stevenson KE, Kehoe SM, Garraway LA, Hahn WC, Meyerson M, Fleming MD, Rollins BJ. Recurrent BRAF mutations in Langerhans cell histiocytosis. Blood. 2010 Sep 16;116(11):1919-23. doi: 10.1182/blood-2010-04-279083. Epub 2010 Jun 2. PMID 20519626
- [Background] Cardoso E, Mercier T, Wagner AD, Homicsko K, Michielin O, Ellefsen-Lavoie K, Cagnon L, Diezi M, Buclin T, Widmer N, Csajka C, Decosterd L. Quantification of the next-generation oral anti-tumor drugs dabrafenib, trametinib, vemurafenib, cobimetinib, pazopanib, regorafenib and two metabolites in human plasma by liquid chromatography-tandem mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2018 Apr 15;1083:124-136. doi: 10.1016/j.jchromb.2018.02.008. Epub 2018 Feb 8. PMID 29544202
- [Background] Donadieu J, Larabi IA, Tardieu M, Visser J, Hutter C, Sieni E, Kabbara N, Barkaoui M, Miron J, Chalard F, Milne P, Haroche J, Cohen F, Helias-Rodzewicz Z, Simon N, Jehanne M, Kolenova A, Pagnier A, Aladjidi N, Schneider P, Plat G, Lutun A, Sonntagbauer A, Lehrnbecher T, Ferster A, Efremova V, Ahlmann M, Blanc L, Nicholson J, Lambilliote A, Boudiaf H, Lissat A, Svojgr K, Bernard F, Elitzur S, Golan M, Evseev D, Maschan M, Idbaih A, Slater O, Minkov M, Taly V, Collin M, Alvarez JC, Emile JF, Heritier S. Vemurafenib for Refractory Multisystem Langerhans Cell Histiocytosis in Children: An International Observational Study. J Clin Oncol. 2019 Nov 1;37(31):2857-2865. doi: 10.1200/JCO.19.00456. Epub 2019 Sep 12. PMID 31513482
- [Background] Haroche J, Cohen-Aubart F, Emile JF, Arnaud L, Maksud P, Charlotte F, Cluzel P, Drier A, Hervier B, Benameur N, Besnard S, Donadieu J, Amoura Z. Dramatic efficacy of vemurafenib in both multisystemic and refractory Erdheim-Chester disease and Langerhans cell histiocytosis harboring the BRAF V600E mutation. Blood. 2013 Feb 28;121(9):1495-500. doi: 10.1182/blood-2012-07-446286. Epub 2012 Dec 20. PMID 23258922
- [Background] Haroche J, Cohen-Aubart F, Emile JF, Donadieu J, Amoura Z. Vemurafenib as first line therapy in BRAF-mutated Langerhans cell histiocytosis. J Am Acad Dermatol. 2015 Jul;73(1):e29-30. doi: 10.1016/j.jaad.2014.10.045. No abstract available. PMID 26089069
- [Background] Heisig A, Sorensen J, Zimmermann SY, Schoning S, Schwabe D, Kvasnicka HM, Schwentner R, Hutter C, Lehrnbecher T. Vemurafenib in Langerhans cell histiocytosis: report of a pediatric patient and review of the literature. Oncotarget. 2018 Apr 24;9(31):22236-22240. doi: 10.18632/oncotarget.25277. eCollection 2018 Apr 24. PMID 29774135
- [Background] Herbrink M, de Vries N, Rosing H, Huitema ADR, Nuijen B, Schellens JHM, Beijnen JH. Development and validation of a liquid chromatography-tandem mass spectrometry analytical method for the therapeutic drug monitoring of eight novel anticancer drugs. Biomed Chromatogr. 2018 Apr;32(4). doi: 10.1002/bmc.4147. Epub 2017 Dec 19. PMID 29165815
- [Background] Heritier S, Jehanne M, Leverger G, Emile JF, Alvarez JC, Haroche J, Donadieu J. Vemurafenib Use in an Infant for High-Risk Langerhans Cell Histiocytosis. JAMA Oncol. 2015 Sep;1(6):836-8. doi: 10.1001/jamaoncol.2015.0736. No abstract available. PMID 26180941
- [Background] Raciborska A, Malas Z, Tysarowski A. [Vemurafenib in refractory langerhans histiocytosis]. Dev Period Med. 2018;22(4):376-378. doi: 10.34763/devperiodmed.20182204.376378. Polish. PMID 30636236
- [Background] Szmulewitz RZ, Ratain MJ. Vemurafenib oral bioavailability: an insoluble problem. J Clin Pharmacol. 2014 Apr;54(4):375-7. doi: 10.1002/jcph.277. No abstract available. PMID 24757719
- [Background] Vikingsson S, Stromqvist M, Svedberg A, Hansson J, Hoiom V, Green H. Novel rapid liquid chromatography tandem masspectrometry method for vemurafenib and metabolites in human plasma, including metabolite concentrations at steady state. Biomed Chromatogr. 2016 Aug;30(8):1234-9. doi: 10.1002/bmc.3672. Epub 2016 Jan 25. PMID 26683023
- [Background] Zhang W, Heinzmann D, Grippo JF. Clinical Pharmacokinetics of Vemurafenib. Clin Pharmacokinet. 2017 Sep;56(9):1033-1043. doi: 10.1007/s40262-017-0523-7. PMID 28255850